CLINICAL TRIAL: NCT05304819
Title: Post-market Clinical Follow-up (PMCF) Study of the AchilloCordPLUS System Implant Set for Acute Achilles Tendon Repair
Brief Title: PMCF Study of the AchilloCordPLUS System Implant Set for Acute Achilles Tendon Repair
Status: Active, not recruiting | Type: Observational
Sponsor: Xiros Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CRE 029
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Achilles Tendon Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- AchilloCordPLUS: End to end repair for acute Achilles tendon rupture with AchilloCordPLUS
  Interventions: Device: AchilloCordPLUS™ System Implant

INTERVENTIONS:
Device: AchilloCordPLUS™ System Implant — AchilloCordPLUS System Implant Set for Acute Achilles Tendon Repair

SUMMARY:
This is a Post Market Clinical Follow Up Study in Orthopaedics, it will verify the long-term safety and performance of the device in the intended patient population, when indicated for the acute repair of the Achilles tendon.

The Medical Device in this study AchilloCordPLUS is a Class IIb UKCA-Marked device manufactured by Xiros Ltd.

DETAILED DESCRIPTION:
This is a Post Market Clinical Follow Up Study in Orthopaedics, it will verify the long-term safety and performance of the device in the intended patient population, when indicated for the acute repair of the Achilles tendon.

The Medical Device in this study AchilloCordPLUS is a Class IIb UKCA-Marked device manufactured by Xiros Ltd.

AchilloCordPLUS is a single-use device, indicated for patients with acute Achilles tendon ruptures. It is particularly suited to active patients where an extended period of postoperative immobilisation is undesirable.

This study is a prospective, single-centre, consecutively recruited non-randomised study. The total length of the study is expected to be 3 years. This includes a recruitment period of approximately 12 months and a 2-year follow-up.

This study has now closed to follow-up, with a recruitment of 19 participants. Follow up is at 2,4,6,8 and 12 weeks, 6 months and 1 and 2 years. All subjects treated with the AchilloCordPLUS for acute Achilles tendon repair will be consecutively recruited into the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be skeletally mature and be 18 years old or above.
* Patients requiring end to end repair for acute Achilles tendon rupture.
* Patient is willing to participate in the study and have been informed of the nature of the study, agree to its follow-up and has provided written informed consent as approved by the Research Ethics Committee (REC).

Exclusion Criteria:

* Patients with chronic ruptures of the Achilles tendon.
* Patients with bilateral ruptures.
* Patients with known hypersensitivity to implant materials. Appropriate tests should be carried out on patients with suspected material sensitivity prior to implantation.
* Patients with infections or any structural or pathological condition of the bone or soft tissue that would be expected to impair healing or prevent secure fixation.
* Patients who are unable or unwilling to restrict activities to prescribed levels or to follow the rehabilitation instructions during the healing period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring end to end repair for acute Achilles tendon rupture.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Achilles Tendon Rupture Score (ATRS) | 6 months
  Change in ATRS Score 0-100 0=major limitations 100=no limitations
adverse events (AE) | 6 months
  Number of adverse events (AE) at 6 months after surgery which directly relate to the procedure that may have an effect on the patient's outcome (for example, irritation at the surgery site, re-rupture, deep-vein thrombosis (DVT), wound infection and sural nerve damage).

SECONDARY OUTCOMES:
Achilles Tendon Rupture Score (ATRS) | 2 years
  Change ATRS Score from baseline upto 2 years in 0-100 0=major limitations 100=no limitations
Length of time to unaided full weight bearing | 2 years
  Length of time to defined as removal of heel raise and walking unaided
return to work and return to sport. | 2 years
  Time for patients to return to work and return to sport.
Tegner Activity Scale (pre-injury) | 2 years
  Number of patients who have returned to pre-injury levels of activity assessed using the Tegner Activity Scale 10 (competitive sport) 0 (sick leave or disability pension)
RAND Short Form 36 (SF 36) V1 | 2 years
  Change from RAND SF 36 Patient-reported quality of life 0-100 a higher sore indicates a higher health state
Tegner Activity Scale (baseline) | 2 years
  Change from Tegner score from baseline to 2 years 10 (competitive sport) 0 (sick leave or disability pension)
Range of Motion | 6 months
  Change in ROM (ankle dorsi and plantar flexion) between each time point up to 6 months after surgery and compare to the contralateral side.
Calf Circumference | 6 months
  Change in calf circumference from 6 weeks up to 6 months and compare to the contralateral side.
Adverse Event | 2 years
  Adverse events up to 2 years after surgery which directly relate to the procedure that may have an effect on the patient's outcome (for example, irritation at the surgery site, rerupture, DVT, wound infection and sural nerve damage).

CONTACTS AND LOCATIONS:
Locations (1):
- North Cumbria Integrated Care Nhs Foundation Trust, Penrith, United Kingdom

IPD SHARING:
Plan to Share IPD: No